CLINICAL TRIAL: NCT01335334
Title: Helicobacter Pylori Eradication Using a Bismuth Quadruple Therapy Among Asymptomatically Infected Adults in El Paso, Texas: A Pilot Study.
Brief Title: H. Pylori Eradication Using Pyklear in Adults in El Paso, Texas: a Pilot Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Victor M. Cardenas, UT HSC School of Public Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UTHSCSPH100386
Record Dates: First submitted 2011-04-12; First posted 2011-04-14 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2011-04

CONDITIONS: H. Pylori Infection
Keywords: Effectiveness; eradication; Asymptomatic
MeSH Terms: interventions — Metronidazole; Tetracycline; Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: bismuth subcitrate potassium, metronidazole,tetracycline hydrochloride and omeprazole — Pylera capsule contains bismuth subcitrate potassium, 140 mg (q.i.d.), metronidazole, 125mg (q.i.d.), tetracycline hydrochloride, 125mg (q.i.d.). Generic omeprazole (20mg, b.i.d) tablets
  Other Names: Pylera; Omeprazole

SUMMARY:
The proposed open-label one arm before-after clinical trial will assess the efficacy of a 14-day quadruple therapy containing 420mg of bismuth subcitrate potassium, 375mg of metronidazole, 375mg of tetracycline hydrochloride (Pylera® packs from Axcan Pharma) and 20mg of omeprazole in eradicating H. pylori infection in 50 asymptomatic adults in El Paso, Texas. As part of the study we will obtain specimens for culture of H. pylori in a reference laboratory.

DETAILED DESCRIPTION:
This study will assess whether this FDA approved treatment taken for 14-days is at least 85% effective in eradicating H. pylori infection.

The study participants will be

* Adults ages 18-65 years
* Able to and who provide written informed consent
* Who meet the inclusion and inclusion criteria

Females of Reproductive Potential

If a female subject becomes pregnant while on this study, the study drug will be discontinued immediately and the subject followed until the outcome of the pregnancy is known. If a pregnancy occurs, it will be reported as an unexpected AE.

Premature Subject Discontinuation

A subject may be discontinued from the study for the following medical or administrative reasons:

* occurrence of an AE, which in the judgment of the investigator suggests an unacceptable risk to the subject (The investigator will follow the subject until satisfactory resolution of the AE or the AE is determined to be stable.);
* development on-study of any condition fulfilling one of the exclusion criteria;
* pregnancy; and/or
* subject request.

The investigator may discontinue individual subjects from the study at any time.

Subjects will be encouraged to complete the study; however they may voluntarily withdraw at any time. The investigator must provide written documentation of the reason for discontinuation on the appropriate study form. Regardless of the reason for or source of withdrawal, all subjects will be asked to undergo an end of therapy evaluation and a 45+-day after completing the study medication. Additionally, subjects who discontinue study drug for any reason, without meeting any of the criteria listed above, may continue in the study. Such subjects will have no further efficacy evaluations following the last study drug dose, but will continue all safety assessments through the 10 days of follow-up. Subjects who withdraw or are withdrawn will not be replaced under this protocol.

Procedures:

* Screening for Helicobacter pylori infection

The investigators will use a novel antibody immunoassay test to detect H. pylori antibodies in urine specimens will be used. The urine sample (0.5 mL) for the RAPIRUN H. pylori antibody test was transferred into a sample diluent tube and will be mixed with the aid of disposable pipette. Approximately 0.2 mL of this mixture will be dropped onto the test device. The test will be considered positive if a colored line is seen in both the test and control windows.

* Confirmation of Helicobacter pylori infection status

For UBT, breath samples will be collected at a visit scheduled 45+ after the end of the eradication treatment, in disposable bags with a one-way valve designed for the use of the UBit 300 (Meretek Diagnostics, LaFayette, CO). A baseline breath sample will be collected at the start of the interview then the subject will be given 150 ml of a drink containing citric acid and 75 mg of 13C-urea. After 20 minutes, a second breath bag will be collected.

* Culture of Helicobacter pylori

Baylor brush cutoffs will be place in 1 ml of cysteine transport medium with 20% glycerol and stored at -70 C until processed at the Laboratory of co-I Dr. Graham where will be cultured in medium consisting of of a horse blood agar (HBA) plate (nonselective medium) or an HBA plate containing 10 μg/ml nalidixic acid, 5 μg/ml trimethoprim, 3 μg/ml, vancomycin and 2 μg/ml amphotericin B (selective medium). MIC testing for clarithromycin, tinidazole and amoxicillin will be conducted using agar dilution methods.

* Screening for Eligibility, pregnancy testing and physical evaluation

Subjects who tested positive to a screening urine test, and subsequently to a urea breath test, will be invited to a visit where the aims, procedures, risks, benefits, and issues of confidentiality and subject's right will be revisited and a consent form will be given for them to take home and review. Subjects will be asked questions to screen for eligibility prior to a clinical evaluation by the Medical director, and will be asked about current medical conditions, dyspepsia symptoms, if currently pregnant, medical personal and family history, and their weight, height, 3' resting blood pressure, heart beat, and temperature will be measured and recorded, a blood sample will be collected to screen for kidney and liver conditions. If the research assistant deems the persons eligible, and willing to take part s/he will schedule an appointment to be seen by Dr. Salazar and bring the signed consent. Subjects will be asked to be fasting for at least eight hours. Once the results of kidney and liver functions are available, the subjects will be seen by Dr. Salazar to assess inclusion and exclusion criteria. At that time, while subjects have been fasting for at least 3 hours, Dr. Salazar will collect samples for culture from gastric mucosa using the Baylor oro-gastric brush as follows: after topical oral anesthesia, the brush assembly is swallowed, the brush is extended in the stomach and to and fro for 3-4 cm, 3-4 times and then retracted into the protective sleeve and withdrawn from the patient (total time after anesthesia ~1 min). The brush will be gently touched to a glass slide for Gram staining, then tip of the brush will be cut off and the brush shaken in a dram vial containing approximately 1 mL of cysteine transport media with 20% glycerol.

* Study medication, dosing and dispensation

Patients will be given a 14-day quadruple [omeprazole (20 mg twice daily) + (420 mg of bismuth subcitrate potassium four times a day)+metronidazole (375 mg four times a day)+ tetracycline hydrochloride (375 mg four times a day) for 14 days.

Each subject will be given 14 daily dosing packs containing 12 PYLERA™ capsules and 2 omeprazole tablets each along with oral and written instructions. Subjects will be asked to repeat the instructions back.

* Follow-up evaluation

A phone call or household visit will take place at day 7. Subjects will be asked "Do you have any new symptom since you started taking the study medication?" Closed-ended question will also ask for solicited adverse events. Also during this evaluation, the study subjects will be asked to provide us with any unused drugs to count the number of tablets and capsules left and record in the appropriate forms. Another visit will be scheduled at day 14 following the same protocol.

* 45+day Evaluation 3 At day 45+ during the sixth visit and will serve the purpose of asking the same question ("Do you have any new symptom since you started taking the study medication?"), collect specimens for a second urea breath test, and complete an exit survey to assess subject's satisfaction with the research experience and obtain their guess of the arm they were assigned to. The validated dyspepsia questionnaire will be administered again to assess changes in symptoms as well.

ELIGIBILITY:
Inclusion Criteria:

* An Institutional Review Board (IRB) approved informed consent is signed and dated prior to any study-related activities.
* Subject is male or female.

If the subject is female, she would be eligible to enter if she is of: Non-childbearing potential (ie, physiologically incapable of becoming pregnant, including any female who has undergone sterilization [hysterectomy or bilateral tubal ligation] or is post-menopausal. For purposes of this study, postmenopausal is defined as 1 year without menses. Women of childbearing potential should have a negative urine pregnancy test at screening and, if heterosexually active, should agree to use a medically approved method of birth control. Medically approved methods of birth control include:

* Double barrier method of contraception, specifically, use of a condom and spermicide, for 1 week prior to study drug administration, throughout the 14 days of treatment and the 7-day follow-up.
* Approved hormonal contraceptives administered for at least 2 monthly cycles prior to study drug administration, throughout the study period and for 1 monthly cycle following completion of study. An intrauterine device (IUD), inserted by a qualified clinician, at least 1 month prior to study drug administration, throughout the study period and for 1 month following completion of the study.
* Partner has undergone vasectomy and subject is in a monogamous relationship.
* Complete abstinence from intercourse for at least 2 weeks prior to study drug administration and throughout the 14-day of treatment. The investigator is responsible for determining whether the subject has adequate birth control for study participation.

  * Subject is at least 18 years of age and not older than 65 years.
  * Subject is infected with H. pylori according to results of a urine antibody test and subsequently confirmed by urea breath testing.
  * Subject is otherwise in good health, free of liver and kidney disease (as determined by medical history and confirmed by liver and kidney tests at baseline).
  * Subject has not received any H. pylori eradication treatment before, not having received antibiotics in the preceding 30 days, or use bismuth compounds more than 3 times per week or other antacids 30 days before taking part in the study.
  * Subject is capable of and willing to comply with all study procedures.

Exclusion Criteria:

* Self-prescribed use of antibiotics, or recent (less than 3 months) of medically prescribed antibiotic treatment for H. pylori eradication.
* Subject is taking a macrolide, amoxicillin, metronidazole or any other imidazole during the study.
* Subject is taking another proton pump inhibitor within 7 days of enrollment unless medically prescribed.
* Subject has hypersensitivity or allergy to penicillin, macrolides or initromidazoles.
* Subject has known or suspected alcohol abuse or illicit drug use within 1 year of enrollment.
* Subject has participated in an investigational drug or device study within the 30 days prior to randomization.
* Subject has concomitant disease or condition that could interfere with, or for which treatment could interfere with the conduct of the study, or could in the opinion of the investigator increase the risk of AEs for the subject's participation in the study, such as having neuropathies or being medically diagnosed with epilepsy.
* Subject is unwilling or unable to comply with the study protocol for any other reason.
* Subject is an alcoholic, according to CAGE questionnaire.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-06 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
H. pylori eradication | 45+ days after treatment
  <2.4 per mil delta over baseline on a urea breath test

CONTACTS AND LOCATIONS:
Locations (1):
- Victor M. Cardenas, El Paso, Texas, United States